CLINICAL TRIAL: NCT04662970
Title: Optimization of Cardiac Resynchronization Therapy by Non-Invasive Imaging of Cardiac Electrophysiology: A Pilot Study
Brief Title: Optimization of Cardiac Resynchronization Therapy by Non-Invasive Imaging of Cardiac Electrophysiology
Acronym: NICE CRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Version 1.2, 09.07.2019
Record Dates: First submitted 2020-11-30; First posted 2020-12-10 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Device programming (Experimental): according to different settings from the SyncAV algorithm
  Interventions: Device: Device programming

INTERVENTIONS:
Device: Device programming — Non-invasive electrophysiology with 65 ECG leads will be performed in 16 different device programming

SUMMARY:
The principal aim is to analyze total left and right ventricular activation time in different CRT device programming algorithms (SyncAV) measured by non-invasive electrophysiology

DETAILED DESCRIPTION:
Patient specific anatomic parameters taken from the cardiac magnetic resonance examination will be the base for a semiautomatic model incorporating the conductivity of the heart, the lungs, blood and the torso. For this reason, a software package (AMIRA Developer, TGS Template Graphics Software, France) has been adapted to calculate a quasi static approximation of Maxwell equations.

After fusion of the T1 CMR scan and the ECG electrodes a model-based bidomain FEM is used for a step-wise measurement of the local activation times (resting potential: 290 mV; plateau: 0 mV; acceleration time: 3 ms) both Ende- and epicardially.

ELIGIBILITY:
Inclusion Criteria:

* patients after successful implantation of a CRT-D or CRT-P device in whom a cardiac magnetic resonance examination is possible and the device is equipped with the SyncAV® programming software
* left bundle branch block before CRT implantation
* PQ interval ≤ 250 ms before implantation

Exclusion Criteria:

* high-grade AV block
* any contraindication concerning a safe CMR performance including claustrophobia
* terminal heart failure (NYHA IV) or cardiac decompensation
* life expectancy < 1 year
* women with child-bearing potential, pregnancy
* drug abusus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Optimal (shortest) activation time of the right and left ventricular in heart failure patients after CRT implantation | The measurements will be done at Day 1
  The activation time will be measured in 16 different device programming settings

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Dichtl, MD PhD, Principal Investigator — Medical University Innsbruck
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No